CLINICAL TRIAL: NCT00014677
Title: A Randomized, Dose-Ranging, Safety and Tolerability Study of NBI-3001 Administered by Continuous Intratumoral Infusion Followed by Surgical Resection in Patients With Recurrent Glioblastoma Multiforme
Brief Title: NBI-3001 Followed by Surgery in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: NBI-3001-0001; CDR0000068586 (Registry Identifier: PDQ (Physician Data Query)); NBI-BB-IND-7004; SLUMC-11350
Record Dates: First submitted 2001-04-10; First posted 2003-11-13 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2002-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — interleukin-4-Pseudomonas exotoxin

INTERVENTIONS:
Biological: interleukin-4 PE38KDEL cytotoxin
Procedure: conventional surgery

SUMMARY:
RATIONALE: NBI-3001 may be able to locate cancer cells and stop them from growing. This may be an effective treatment for glioblastoma multiforme.

PURPOSE: Randomized phase II trial to compare different regimens of NBI-3001 followed by surgery to remove the tumor in treating patients who have glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety, tolerability, and optimal clinical dose of interleukin-4(38-37)-PE38KDEL cytotoxin (NBI-3001) followed by surgical resection in patients with recurrent glioblastoma multiforme.

OUTLINE: This is an open-label, dose-escalation, multicenter study. Patients receive interleukin-4(38-37)-PE38KDEL cytotoxin (NBI-3001) intratumorally as a continuous infusion over 4-5 days beginning within 12-36 hours after ventricular catheter placement. Patients then undergo surgical tumor resection approximately 3 weeks after drug infusion. Cohorts of 6 patients receive escalating doses of NBI-3001 until the maximum tolerated dose is determined. Patients are followed within 1 week and then at 8, 16, and 26 weeks.

PROJECTED ACCRUAL: Approximately 30-36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or progressive glioblastoma multiforme Previously treated with cytoreductive surgery Unilateral, unifocal tumor with a volume of 5-80 mL Not eligible for further radiotherapy due to prior external beam radiotherapy No multifocal, brain stem, or infratentorial tumor or tumor invading midline No tumor with a clinically significant mass effect (greater than 5 mm midline shift) while on stable dose of corticosteroid No clinical symptoms attributed to uncontrolled increased intracranial pressure and/or edema of the brain

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No focal or generalized seizure(s) within 30 days prior to enrollment No other prior or concurrent malignancy except carcinoma in situ of the cervix or basal cell or squamous cell skin cancer No medical instability due to non-malignant systemic disease No other prior or concurrent condition that would preclude study compliance Not pregnant Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior antineoplastic chemotherapy Endocrine therapy: See Disease Characteristics Stable dose of dexamethasone for at least 72 hours prior to catheter placement Radiotherapy: See Disease Characteristics No prior radiosurgery boost (e.g., gamma knife or stereotactic radiosurgery) At least 8 weeks since prior radiotherapy Surgery: See Disease Characteristics At least 4 weeks since prior craniotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Primary Completion 2002-09 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Pan, MD, PhD, Study Chair — Neurocrine Biosciences
Locations (4):
- United States (4):
  - UCSD Thornton Hospital, La Jolla, California
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Charlotte Neurosurgical Associates, Charlotte, North Carolina